CLINICAL TRIAL: NCT03227341
Title: Does Pulmonary Rehabilitation Contribute to Asthma Control?
Brief Title: Pulmonary Rehabilitation in Asthma Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof. Ilknur NAZ, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KCU123
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: asthma control; pulmonary rehabilitation
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with uncontrolled asthma. (Other): 8 week pulmonary rehabilitation program
  Interventions: Other: Exercise
- patients with partially controlled asthma (Other): 8 week pulmonary rehabilitation program
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 8 week exercise program including breathing exercises consisted of pursed-lip breathing, diaphragmatic breathing and thoracic expansion exercises, relaxation and stretching exercises, upper and lower extremity muscle strength training, and aerobic exercises. In addition, bronchial hygiene techniques and dyspnea-reducing positions

SUMMARY:
The investigators compared the effectiveness of pulmonary rehabilitation program on asthma control in patients with uncontrolled and partially controlled asthma.

DETAILED DESCRIPTION:
Asthma treatment is not only medical, it also requires a comprehensive care including nonpharmacological treatment. Pulmonary rehabilitation represents the most important part of the comprehensive care. The investigators aimed to evaluate the efficacy of pulmonary rehabilitation in patients with uncontrolled and partially controlled asthma.

Asthma patients referred to pulmonary rehabilitation (PR) unit were classified according to asthma control test; as partially controlled patients (Group 1), and as uncontrolled patients (Group 2). All patients received of a 8 week pulmonary rehabilitation program. Asthma control tests, pulmonary function tests, arterial blood gases analysis, dyspnea perception, quality of life, exercise capacity, anxiety and depression assessments were performed before and after pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients referred from the outpatient clinic to Pulmonary Rehabilitation unit was confirmed according to GINA guidelines

Exclusion Criteria:

* If the initial diagnosis cannot be confirmed, the patient excluded from the study
* Patients were under medical treatment of -6 months and considered clinically stable.
* Patients with cardiovascular, other lung diseases (pneumoconiosis, pulmonary tuberculosis, interstitial lung disease), or musculoskeletal diseases that would impair exercise training were excluded from the study.
* Also subjects with lack of motivation, poor compliance (not attending the program more than 2 times) or having transport problems were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Asthma control test score | 4 weeks
  A test measured the control of asthma

SECONDARY OUTCOMES:
Exercise capacity | 6 minute
  Six minute walk test
Dyspnea | 1 year
  MMRC Dyspnea Scale
Quality of Life | 1 year
  St. George Respiratory Questionnaire
Pulmonary Function Test | 1 hour
  FEV1, FVC, DLCO
Arterial Blood Gas | 1 hour
  PaO2, PaCO2, SaO2
Anxiety and Depression | 1 week
  Hospital Anxiety and Depression Scale

IPD SHARING:
Plan to Share IPD: Undecided